CLINICAL TRIAL: NCT02720367
Title: A Phase 1b, Multicenter, Open Label Study Evaluating Safety, Tolerability and Preliminary Efficacy of GemRIS 225 mg in Subjects With Non-Muscle-Invasive Urothelial Carcinoma of the Bladder
Brief Title: Safety and Tolerability of TAR-200 mg in Subjects With Non-Muscle-Invasive Bladder Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taris Biomedical LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAR-200-102; 2016-000099-66 (EudraCT Number)
Record Dates: First submitted 2016-02-25; First posted 2016-03-25 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Urinary Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 7-Day Regimen (Experimental): TAR-200 is placed into the bladder through an inserter on Study Day 0 and is removed on Study Day 7. TAR-200 releases gemcitabine gradually during the 7 day indwelling time. A second TAR-200 is placed in the bladder on Study Day 21 and is removed on Study Day 28, which is the day of the TURBT.
  Interventions: Drug: Gemcitabine-Releasing Intravesical System (GemRIS)/TAR-200
- 21-Day Regimen (Experimental): TAR-200 is placed into the bladder through an inserter on Study Day 0 and is removed on Study Day 21. TAR-200 releases gemcitabine gradually during the 21 day indwelling time. A second TAR-200 is placed in the bladder on Study Day 21 and is removed on Study Day 42.
  Interventions: Drug: Gemcitabine-Releasing Intravesical System (GemRIS)/TAR-200

INTERVENTIONS:
Drug: Gemcitabine-Releasing Intravesical System (GemRIS)/TAR-200 — TAR-200 is a passive, nonresorbable gemcitabine-releasing intravesical system whose primary mode of action is the controlled release of gemcitabine into the bladder over an indwelling period.

SUMMARY:
The purpose of this study is to determine if TAR-200, an investigational drug-delivery system is safe and tolerable in patients with recurrent low or intermediate risk non-muscle-invasive bladder cancer (NMIBC) between diagnosis and transurethral resection of bladder tumors (TURBT)

ELIGIBILITY:
Inclusion Criteria:

* A documented history of histologically-confirmed low or intermediate risk urothelial carcinoma of the bladder, excluding carcinoma in situ (pTis), pathologic stage pT1 (invasive into lamina propria) and high-Grade disease, judged not to be muscle infiltrating (pT2 or greater) and accessible for resection.
* Adequate laboratory parameters.
* Screening urinalysis showing no clinically significant abnormalities except those attributable to bladder cancer.
* Not undergoing active treatment in last 3 months for prior or concurrent neoplastic disease and have fully recovered from treatment effects. Patients undergoing concurrent hormonal therapy treatment for prostate cancer will be allowed to enroll.

Exclusion Criteria:

* Exposure to BCG therapy and/or any other intravesical. chemotherapeutic agent less than 1 year prior to enrollment, except single postoperative instillations.
* Absence of visible tumor at Screening.
* Any previous exposure to intravesical gemcitabine instillations within the past 12 months.
* Presence of any bladder or urethral anatomical feature that in the opinion of the investigator may prevent the safe placement, indwelling use or removal of TAR-200 (i.e. bladder diverticula, complete incontinence).
* Patients with a high-Grade urine cytology at recurrence.
* Currently receiving other systemic or intravesical chemotherapy.
* Pelvic radiotherapy administered within 6 months prior to enrollment. Patients who received radiotherapy ≥ 6 months prior to enrollment must demonstrate no cystoscopic evidence or clinical symptoms of radiation cystitis.
* Bladder Post-Void Residual Volume (PVR) of > 250-mL.
* Active, uncontrolled urogenital bacterial, viral, or fungal infections, including urinary tract infection. Skin/nail fungal infections are not exclusionary. Subjects with active shingles (varicella zoster infection) will be excluded from the study.
* History or presence of any significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, gynecological, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder that, in the opinion of the investigator, contraindicates participation.
* Concomitant immunosuppressive medications, such as methotrexate or TNF inhibitors, within 2 weeks of Study Day 0, exclusive of steroid doses ≤5 mg daily.
* Female subject who is pregnant (as verified by urine test at time of screening) or lactating, or of childbearing potential and not using acceptable methods of contraception.
* Unwilling or unable to provide informed consent or comply with the requirements of this protocol, including the presence of any condition (physical, mental or social) that is likely to affect the subject's return for scheduled visits and follow-up.
* Other unspecified reasons that, in the opinion of the investigator or TARIS, make the patient unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Safety as defined by the number of participants with treatment emergent adverse events (TEAEs) coded with MedDRA and graded for severity with CTCAE v4.0 | From the point of signing the informed consent form through last study visit, up to 59 days.

SECONDARY OUTCOMES:
Number of participants who are tolerant of TAR-200 indwelling (Arm 1) | From Day 0 up to Day 7
Percentage of participants who are tolerant of TAR-200 indwelling (Arm 1) | From Day 0 up to Day 7
Number of participants who are tolerant of TAR-200 indwelling (Arm 1) | From Day 21 up to Day 28
Percentage of participants who are tolerant of TAR-200 indwelling (Arm 1) | From Day 21 up to Day 28
Cmax, plasma dFdU (Arm 1) | From Day 0 up to Day 32
  Analysis of Cmax (maximum concentration achieved over time) of diflourodeoxyuridine (dFdU) in plasma.
Tmax, plasma dFdU (Arm 1) | From Day 0 up to Day 32
  Analysis of Tmax (Day at which maximum concentration was achieved) of diflourodeoxyuridine (dFdU) in plasma.
Cavg, plasma dFdU (Arm 1) | From Day 0 up to Day 32
  Analysis of Descriptive statistics (e.g. sample size, mean and median, quartiles, minimum and maximum and box plots) of the concentration of diflourodeoxyuridine (dFdU) in plasma.
Cmax, plasma dFdC (Arm 1) | From Day 0 up to Day 32
  Analysis of Cmax (maximum concentration achieved over time) of gemcitabine (deoxydifluorocytidine hydrochloride - dFdC) in plasma.
Tmax, plasma dFdC (Arm 1) | From Day 0 up to Day 32
  Analysis of Tmax (Day at which maximum concentration was achieved) of gemcitabine (deoxydifluorocytidine hydrochloride - dFdC) in plasma
Cavg, plasma dFdC (Arm 1) | From Day 0 up to Day 32
  Analysis of Descriptive statistics (e.g. sample size, mean and median, quartiles, minimum and maximum and box plots) of the concentration of gemcitabine (deoxydifluorocytidine hydrochloride - dFdC) in plasma.
Cmax, urine dFdU (Arm 1) | From Day 0 up to Day 32
  Analysis of Cmax (maximum concentration achieved over time) of diflourodeoxyuridine (dFdU) in urine.
Tmax, urine dFdU (Arm 1) | From Day 0 up to Day 32
  Analysis of Tmax (Day at which maximum concentration was achieved) of diflourodeoxyuridine (dFdU) in urine
Cavg, urine dFdU (Arm 1) | From Day 0 up to Day 32
  Analysis of Descriptive statistics (e.g. sample size, mean and median, quartiles, minimum and maximum and box plots) of the concentration of diflourodeoxyuridine (dFdU) in urine.
Cmax, urine dFdC (Arm 1) | From Day 0 up to Day 32
  Analysis of Cmax (maximum concentration achieved over time) of gemcitabine (deoxydifluorocytidine hydrochloride - dFdC) in urine.
Tmax, urine dFdC (Arm 1) | From Day 0 up to Day 32
  Analysis of Tmax (Day at which maximum concentration was achieved) of gemcitabine (deoxydifluorocytidine hydrochloride - dFdC) in urine.
Cavg, urine dFdC (Arm 1) | From Day 0 up to Day 32
  Analysis of Descriptive statistics (e.g. sample size, mean and median, quartiles, minimum and maximum and box plots) of the concentration of gemcitabine (deoxydifluorocytidine hydrochloride - dFdC) in urine
Preliminary anti-tumor effects will be assessed in tumor material (post-treatment) for assessment of immunohistochemical tissue biomarkers of drug-induced cell death (AKT, CD31, Ki67, TUNEL). (Arm 1) | Anti-tumor analysis will occur at the following study day visit Day 28
Number of participants who are tolerant of TAR-200 indwelling (Arm 2) | From Day 0 up to Day 21
Percentage of participants who are tolerant of TAR-200 indwelling (Arm 2) | From Day 0 up to Day 21
Number of participants who are tolerant of TAR-200 indwelling (Arm 2) | From Day 21 up to Day 42
Percentage of participants who are tolerant of TAR-200 indwelling (Arm 2) | From Day 21 up to Day 42
Cmax, plasma dFdU (Arm 2) | From Day 0 up to Day 47
  Analysis of Cmax (maximum concentration achieved over time) of diflourodeoxyuridine (dFdU) in plasma.
Tmax, plasma dFdU (Arm 2) | From Day 0 up to Day 47
  Analysis of Tmax (Day at which maximum concentration was achieved) of diflourodeoxyuridine (dFdU) in plasma.
Cavg, plasma dFdU (Arm 2) | From Day 0 up to Day 47
  Analysis of Descriptive statistics (e.g. sample size, mean and median, quartiles, minimum and maximum and box plots) of the concentration of diflourodeoxyuridine (dFdU) in plasma.
Cmax, plasma dFdC (Arm 2) | From Day 0 up to Day 47
  Analysis of Cmax (maximum concentration achieved over time) of gemcitabine (deoxydifluorocytidine hydrochloride - dFdC) in plasma.
Tmax, plasma dFdC (Arm 2) | From Day 0 up to Day 47
  Analysis of Tmax (Day at which maximum concentration was achieved) of gemcitabine (deoxydifluorocytidine hydrochloride - dFdC) in plasma
Cavg, plasma dFdC (Arm 2) | From Day 0 up to Day 47
  Analysis of Descriptive statistics (e.g. sample size, mean and median, quartiles, minimum and maximum and box plots) of the concentration of gemcitabine (deoxydifluorocytidine hydrochloride - dFdC) in plasma.
Cmax, urine dFdU (Arm 2) | From Day 0 up to Day 47
  Analysis of Cmax (maximum concentration achieved over time) of diflourodeoxyuridine (dFdU) in urine.
Tmax, urine dFdU (Arm 2) | From Day 0 up to Day 47
  Analysis of Tmax (Day at which maximum concentration was achieved) of diflourodeoxyuridine (dFdU) in urine
Cavg, urine dFdU (Arm 2) | From Day 0 up to Day 47
  Analysis of Descriptive statistics (e.g. sample size, mean and median, quartiles, minimum and maximum and box plots) of the concentration of diflourodeoxyuridine (dFdU) in urine.
Cmax, urine dFdC (Arm 2) | From Day 0 up to Day 47
  Analysis of Cmax (maximum concentration achieved over time) of gemcitabine (deoxydifluorocytidine hydrochloride - dFdC) in urine.
Tmax, urine dFdC (Arm 2) | From Day 0 up to Day 47
  Analysis of Tmax (Day at which maximum concentration was achieved) of gemcitabine (deoxydifluorocytidine hydrochloride - dFdC) in urine.
Cavg, urine dFdC (Arm 2) | From Day 0 up to Day 47
  Analysis of Descriptive statistics (e.g. sample size, mean and median, quartiles, minimum and maximum and box plots) of the concentration of gemcitabine (deoxydifluorocytidine hydrochloride - dFdC) in urine
Preliminary anti-tumor effects will be assessed in tumor material (post-treatment) for assessment of immunohistochemical tissue biomarkers of drug-induced cell death (AKT, CD31, Ki67, TUNEL). (Arm 2) | Anti-tumor analysis will occur at the following study day visit Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Witjes, MD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Radboudumc, Nijmegen